CLINICAL TRIAL: NCT03797950
Title: Mobile Nudges to Increase Early Vaccination Coverage in Rural Areas: A Pilot Investigation in Ghana's Northern Region
Brief Title: Mobile Nudges to Increase Early Vaccination Coverage in Rural Areas
Acronym: GEVaP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Tropical & Public Health Institute (Other)
Collaborators: Innovations for Poverty Action (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: GHS-ERC008/07/18
Record Dates: First submitted 2018-11-07; First posted 2019-01-09 (Actual); Last update posted 2020-03-03 (Actual); Status verified 2020-03

CONDITIONS: Immunization Coverage
Keywords: OPV; BCG; vaccine delivery; mhealth; incentives

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): No active intervention
- Voice Reminder (Group A) (Experimental): Community-appointed volunteers will document births in the community and will receive small monetary rewards via "mobile money" for all documented births. Enrolled women will receive reminders via mobile phone to highlight the importance of early vaccinations for newborns. Messages will recommend that women take their newborns to get the BCG and Polio0 vaccine as soon as possible after birth (within the first two weeks of life for Polio0 and within the first month for BCG). Information on where and when these vaccines will be available in the woman's community will be provided.
  Interventions: Behavioral: Voice Reminder (Group A)
- Cash Incentive (Group B) (Experimental): Community-appointed volunteers will document births in the community and will receive small monetary rewards via "mobile money" for all documented births. Volunteers will encourage enrolled women to seek early vaccination for their newborns. Messages will recommend that women take their newborns to get the BCG and Polio0 vaccine as soon as possible after birth (within the first two weeks of life for Polio0 and within the first month for BCG). Volunteers will provide information on where and when these vaccines will be available in the woman's community. Volunteers and enrolled women will receive small monetary rewards via "mobile money" for receiving OPV0 and BCG vaccinations on time.
  Interventions: Behavioral: Cash Incentive (Group B)

INTERVENTIONS:
Behavioral: Voice Reminder (Group A) — Woman with a recent delivery will be contacted via mobile phone by a central study staff member to encourage them to vaccinate their newborn with OPV0 and BCG, and information on where and when vaccines are available in this community will be provided. Community volunteers will receive small incentives for documenting births in the community.
  Arms: Voice Reminder (Group A)
Behavioral: Cash Incentive (Group B) — Mobile phone based monetary incentives will be provided to community volunteers and to women with a recent delivery who vaccinate newborns with OPV0 and BCG on time. Community volunteers will receive small incentives for documenting births in the community.
  Arms: Cash Incentive (Group B)

SUMMARY:
Despite major progress made in vaccination coverage overall, timeliness of vaccines remains a key concern in many settings. At the same time, access to mobile phones has increased rapidly, offering new opportunities to track and deliver health services. This research project uses these newly available mobile phone networks to simultaneously address two of the biggest bottlenecks in vaccine delivery: timely documentation of births, and lack of maternal effort or access to get essential vaccines. To increase documentation, investigators will train volunteers in each community to report new births via mobile phone to a central coordinator, and send small monetary rewards via mobile phone to volunteers for this reporting. To increase vaccination coverage, investigators will send reminder messages directly to mothers, and will also test small monetary rewards to volunteers and to mothers as an incentive to complete recommended vaccinations. The designs to provide vaccination encouragement will be tested through a small community randomized controlled trial in 15 selected villages in Ghana's Northern region. The primary outcome for the pilot study will be the percentage of children who received both the polio birth dose (OPV0) vaccination within two weeks of life (14 days) and the BCG vaccination within the first four weeks (28 days) of life.

DETAILED DESCRIPTION:
Despite major progress made in vaccination coverage overall, timeliness of vaccines remains a key concern in many settings. Early vaccination coverage is particularly low in settings where a large share of women deliver at home, as it is the case in Ghana's Northern region, where only a minority of women seek out facilities for delivery. In Ghana, 95% of children receive BCG vaccination within the first two years of life, but only about half of these children receive the vaccine within the first 30 days after delivery. Less than 50% of children in Ghana's Northern region receive Bacillus Calmette-Guérin (BCG) vaccines within the first three months of their life, and less than 40% get polio vaccination, exposing a large number of infants to these diseases.

Recent research conducted in this region shows that the large majority of households have access to mobile phones, even in the most rural areas. this project uses mobile phone networks to simultaneously address two of the biggest bottlenecks in vaccine delivery: timely documentation of births, and lack of maternal effort or access to essential vaccines. Evidence from other low resource settings suggests that even small rewards can often result in substantial increases in vaccine uptake - investigators will test this hypothesis using mobile networks in rural areas of Northern Ghana.

The main objective of this study is to assess the extent to which mobile-phone based reminder or reward systems can increase early vaccination coverage. Investigators will assess two specific interventions through the pilot study:

1. a mobile-phone based call and text system which will be used to contact mothers to highlight the importance of early vaccinations, provide reminders (nudges) to mothers encouraging them to get their newborn vaccinated and providing information on where and when vaccinations are available in their community.
2. a community volunteer-based system that will provide small mobile credit rewards to both community volunteers and mothers for completing the early vaccinations within the first month of newborn life.

Research Hypotheses (H1-3) H1: Nudging mothers through voice and text messages will increase early vaccination coverage.

H2: Nudging mothers through community volunteers and small rewards will increase early vaccination coverage.

Given that birth documentation remains low in many parts of Ghana, investigators will also test a new community-based reporting model, under which volunteers appointed by the community will receive small rewards for reporting births that occur in their communities. Investigators will test the extent to which such a program results in successful reporting of births:

H3: Providing small mobile-phone based incentives to volunteers selected by communities for reporting births will result in accurate and timely reporting of births in rural areas.

The study is an open label cluster-randomized controlled trial with three arms: a control arm, a voice reminder arm (group A), and a cash incentive arm (group B). During the intervention phase community volunteers will be appointed to document all births in 10 randomly selected treatment communities (group A and group B), and will receive small cash rewards delivered via "mobile money" for all documented births. In each of two active treatment arms, women across five villages will be enrolled in a proactive program over a period of six months. In intervention group A, participating women will receive reminders about vaccinations recommended at birth delivered via mobile phones. In intervention group B, participating women will receive encouragement from a community-appointed volunteer to complete recommended vaccinations and community volunteers and woman will receive small cash rewards delivered via "mobile money" for completing the recommended birth dose vaccinations on time. No volunteer will be appointed to documents births in the 5 control-arm villages and no women in the 5 control-arm villages will be actively enrolled nor receive a pro-active program intervention during the intervention phase.

After the intervention phase is complete, an endline population-based household survey will be conducted in the 15 study villages (5 control, 5 treatment group A, 5 treatment group B) to evaluate the effect of the intervention programs on vaccine coverage.

ELIGIBILITY:
Inclusion Criteria:

* Women who have given birth to a live-born, surviving infant in the last two weeks (14 days) and reside in the community.

Exclusion Criteria:

* Women who do not reside in the community.
* Women whose newborn has passed away.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Woman who have recently given birth
Enrollment: 260 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-07-09 (Actual); Study Completion 2019-07-09 (Actual)

PRIMARY OUTCOMES:
Full on time early vaccination coverage (OPV0 and BCG) | First month of life
  Percentage of infants born during study who received both BCG and OPV0 vaccinations on time (OPV0 within first 2 weeks of life and BCG within first month of life)

SECONDARY OUTCOMES:
On time BCG coverage | First month of life
  Percentage of infants who received BCG vaccination on time (within first month of life)
On time OPV coverage | First two weeks of life (14 days)
  Percentage of infants born during study who received OPV0 on time (within first two weeks of life)

OTHER OUTCOMES:
Birth documentation and reporting coverage | First month of life
  Percentage of live births in the community during the study which are documented and reported by community health volunteers

CONTACTS AND LOCATIONS:
Overall Officials: Guenther Fink, PhD, Principal Investigator — Swiss Institute for Tropical and Public Health
Locations (1):
- Innovations for Poverty Action, Tamale, Karaga, Ghana

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Levine G, Salifu A, Mohammed I, Fink G. Mobile nudges and financial incentives to improve coverage of timely neonatal vaccination in rural areas (GEVaP trial): A 3-armed cluster randomized controlled trial in Northern Ghana. PLoS One. 2021 May 19;16(5):e0247485. doi: 10.1371/journal.pone.0247485. eCollection 2021. PMID 34010312
- [Derived] Palmer MJ, Henschke N, Bergman H, Villanueva G, Maayan N, Tamrat T, Mehl GL, Glenton C, Lewin S, Fonhus MS, Free C. Targeted client communication via mobile devices for improving maternal, neonatal, and child health. Cochrane Database Syst Rev. 2020 Jul 14;8(8):CD013679. doi: 10.1002/14651858.CD013679. PMID 32813276